CLINICAL TRIAL: NCT07108452
Title: Leveraging AI to Transform Dietary Choices for Cardiovascular Health in Young Adults Experiencing Food Insecurity
Brief Title: Using an AI Mobile Application to Promote Healthy Eating
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: International Food Policy Research Institute (Other); Penn State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2308774; 25ISA1474935 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2025-07-08; First posted 2025-08-07 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Healthy
Keywords: artificial intelligence; Implementation science; college students; food security; diet quality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group- Gamified app version; dietary assessment + gamification (Experimental): Participants will be randomly assigned at enrollment to the intervention group, which will receive a gamified app that delivers behavioral nudges and provides a daily report of caloric and nutrient intake.
  Interventions: Other: A mobile application that uses AI to deliver behavioral nudges that encourage healthy food choices.
- Control group- Limited app version, dietary assessment only (Active Comparator): Participants will be randomized at enrollment to the control group, which will receive a "limited" app version that only provides a daily report of caloric and nutrient intake, without delivering behavioral nudges.
  Interventions: Other: Limited app version for dietary assessment only

INTERVENTIONS:
Other: A mobile application that uses AI to deliver behavioral nudges that encourage healthy food choices. — As a mobile application for assessing dietary intake, the app provides a daily report of food intake- a core function that both the gamified and limited app versions have. The gamified version has the added functionality of delivering behavioral nudges that encourage healthy food selections.
  Arms: Intervention group- Gamified app version; dietary assessment + gamification
Other: Limited app version for dietary assessment only — This app version provides a daily report of energy and nutrient intake- available to those randomized to the control group
  Arms: Control group- Limited app version, dietary assessment only

SUMMARY:
The goal of this feasibility study is to determine the adherence, acceptability, and usability of the behavioral intervention of a mobile AI application and its effects on food choices and diet quality. A secondary goal is to assess whether the app's accuracy or feasibility differs by food security status. Study participants are UC Davis students aged 18-24 years. The main question it aims to answer is:

- Does the gamified app version that delivers behavioral nudges have a higher adherence and acceptability rate, and does this translate to better dietary behaviors?

Participants will use either the intervention app (dietary assessment + gamification) or the control app (non-gamified, dietary assessment only) for six weeks to record all their food intake. Diet quality will be assessed at baseline and endline, and a Likert scale acceptability questionnaire will be administered at endline.

ELIGIBILITY:
Inclusion Criteria:

* Willing to use their smartphones with app to record all foods consumed
* UC Davis student

Exclusion Criteria:

* eating disorders
* Participant in the validation study that tested the app's accuracy against weighed food records

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 114 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
App acceptability by version assigned to participants | Measured at endline: at the end of the 6 week period
  Acceptability will be assessed using a structured questionnaire based on a Likert scale from 1 (strongly agree) to 5 (strongly disagree) administered at the end of the study period.
App's usability by version assigned to participants | Measured at endline: at the end of the 6 week period
  Focus group discussions will be conducted with a select group of participants to assess usability (i.e. facilitators and barriers to app usage) at the end of the study period.
App adherence rates by version assigned to participants | Assessed at midline (3 weeks) and endline (6 weeks)
  App usage adherence will be evaluated based on analytics data, with a 70% usage threshold defined for both the midline and endline assessments.

SECONDARY OUTCOMES:
Diet quality assessment by app version, measured using Healthy Eating Index scores at baseline and endline. | From enrollment till study completion at 6 weeks
  Determine changes in diet quality by app version. The Healthy Eating Index is scored from 0-100. The higher the score, the better the alignment of a diet with key recommendations in the Dietary Guidelines for Americans.
App usability by food security status assessed using the USDA 10-item food security survey module | Food security assessed at baseline
  The validated USDA 10-item Food Security Survey Module will be used to capture food security over the prior 12 months and be administered at the recruitment visit. Moderation of app's usability by food security status will be assessed by including an interaction term between the app version and food security strata. Food security status is assigned as follows- Raw score zero: High food security; Raw score 1-2: Marginal food security; Raw score 3-5: Low food security; Raw score 6-10:Very low food security.
App acceptability by food security status assessed using the USDA 10-item food security survey module | Food security assessed at baseline
  The validated USDA 10-item Food Security Survey Module will be used to capture food security over the prior 12 months and be administered at the recruitment visit. Moderation of app's acceptability by food security status will be assessed by including an interaction term between the app version and food security strata. Food security status is assigned as follows- Raw score zero: High food security; Raw score 1-2: Marginal food security; Raw score 3-5: Low food security; Raw score 6-10:Very low food security.
App adherence rates by food security status assessed using the USDA 10-item food security survey module | Food security assessed at baseline
  The validated USDA 10-item Food Security Survey Module will be used to capture food security over the prior 12 months and be administered at the recruitment visit. Moderation of app's adherence rates by food security status will be assessed by including an interaction term between the app version and food security strata. Food security status is assigned as follows- Raw score zero: High food security; Raw score 1-2: Marginal food security; Raw score 3-5: Low food security; Raw score 6-10:Very low food security.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren E Au, PhD, RDN, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis - Department of Nutrition, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2025-06-04): https://cdn.clinicaltrials.gov/large-docs/52/NCT07108452/Prot_SAP_000.pdf
  • Informed Consent Form: Pilot RCT (2025-06-04): https://cdn.clinicaltrials.gov/large-docs/52/NCT07108452/ICF_001.pdf
  • Informed Consent Form: Validation study (2025-06-04): https://cdn.clinicaltrials.gov/large-docs/52/NCT07108452/ICF_002.pdf